CLINICAL TRIAL: NCT00871273
Title: A Pharmacokinetic Study of Capecitabine in Patients Undergoing Peri-operative Chemotherapy and a Total Gastrectomy for Adenocarcinoma of the Stomach
Brief Title: Pharmacokinetic Study of Capecitabine After Total Gastrectomy for Stomach Adenocarcinoma
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: 1. Slow recruitment; 2. Change to clinical environment reducing the pool of potentially eligible patients; 3. Availability of data from another similar study
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Duncan Jodrell, Professor Duncan Jodrell, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CAP002
Record Dates: First submitted 2009-03-27; First posted 2009-03-30 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Adenocarcinoma of the Stomach
Keywords: capecitabine; total gastrectomy; pharmacokinetic
MeSH Terms: interventions — Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: capecitabine — film-coated tablet 1250 mg/m2 twice daily 14 days for 14 days. Number of cycles: 3 cycles pre-operatively and 3 cycles post-operatively unless there is evidence of disease progression on chemotherapy
  Other Names: Xeloda

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK) of capecitabine in patients who have undergone a total gastrectomy.

DETAILED DESCRIPTION:
Primary Objective:

* To establish the pharmacokinetics (PK) of capecitabine in patients who have undergone a total gastrectomy

Secondary Objectives:

* To compare the pharmacokinetic profile of capecitabine administered to patients with gastric cancer pre- and post-gastrectomy and to compare this to historical data of capecitabine PK values in patients with other cancer types.
* To ensure equivalent capecitabine exposure when compared to PK data from the same patients prior to gastrectomy.

This is a clinical trial to evaluate the pharmacokinetics (PK) of capecitabine in patients who have undergone a total gastrectomy. The study also aims to establish the toxicity profile of capecitabine in these patients, to identify any dose limiting toxicities (DLT), and to ensure equivalent capecitabine exposure when compared to PK data from the same patients prior to gastrectomy. Screening tests will consist of demographic details, complete medical history, physical exam, vital signs, tumour serum markers, haematology and biochemistry tests. There will also be an ECG, chest X-Ray or CT thorax, CT abdomen and a serum or urine pregnancy test (for women of childbearing potential). Haematology and Biochemistry will be repeated prior to each study drug administration. All patients will receive 6 cycles of oral capecitabine chemotherapy at a dose of 625 mg/m2, administered twice daily at 12 hourly intervals for 21 consecutive days. Total proposed duration of therapy is 3 cycles pre-operatively and 3 cycles post-operatively. Capecitabine and its metabolites (DFCR, DFUR and 5-FU) plasma levels will be measured during the 1st and 4th cycles in all patients. Treatment should continue for 6 cycles unless there is evidence of disease progression, or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed gastric carcinoma suitable for potentially curative resection.
* Surgery must be planned to involve a total gastrectomy.
* No concurrent mechanical or malabsorptive disorders precluding affective oral administration of the drug (excluding early satiety related to the presence of the malignancy).
* Age ≥ 18 years.
* World Health Organisation (WHO) performance status of ≤ 2 (Appendix 1).
* Haematological and biochemical indices (These measurements must be performed within one week prior to the patient going on study.)
* Haemoglobin (Hb) ≥ 9.0 g/dl
* Neutrophils ≥ 1.5 x 109/L
* Platelets (Plts) ≥ 100 x 109/L
* Serum bilirubin ≤ 1.5 x upper normal limit
* Alanine amino-transferase (ALT) and / or aspartate amino-transferase (AST) ≤ 2.0 x upper limit of normal (ULN). (If both are measured, both must be ≤ 2.0 x ULN)
* Calculated creatinine clearance ≥ 50 ml/min (uncorrected value) or isotope clearance measurement ≥ 50ml/min
* Female patients of child-bearing potential must have a negative serum or urine pregnancy test prior to enrolment and agree to use appropriate medically approved contraception for four weeks prior to entering the trial, during the trial, and for six months afterwards.
* Male patients must agree to use appropriate medically approved contraception during the trial and for six months afterwards.
* Written, informed consent provided.
* Ability of the patient to co-operate with treatment and follow up must be ensured.
* Patients receiving oral anti-coagulation prior to entry into the study, must be converted to low molecular weight heparin in light of the interaction between capecitabine and warfarin.

Exclusion Criteria:

* Patients with gastric lymphoma or other histological diagnosis
* Any evidence of malignant ascites, peritoneal or liver metastasis, spread to other distant abdominal or extra-abdominal organs.
* History of confirmed Ischaemic Heart Disease, concurrent congestive heart failure or prior history of class III / IV cardiac disease (Appendix 2 - New York Heart Association (NYHA) Scale)
* Concurrent mechanical or malabsorptive disorders precluding effective oral administration of the drug
* Use of other concomitant chemotherapy
* Pregnancy or Lactation
* Patients known to be serologically positive for Hepatitis B, Hepatitis C or Human Immunodeficiency Virus (HIV).
* Patients who are high medical risks because of non-malignant systemic disease including active uncontrolled infection.
* Any other serious medical or psychological condition precluding adjuvant treatment
* Patients with any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-11; Primary Completion 2013-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
To establish the pharmacokinetics (PK) of capecitabine in patients who have undergone a total gastrectomy. | Samples collected predose and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 8, and 24 hours on day 1 of cycles 1 and 4

SECONDARY OUTCOMES:
To compare the pharmacokinetic profile of capecitabine administered to patients with gastric cancer pre- and post-gastrectomy and to compare this to historical data of capecitabine PK values in patients with other cancer types. | 1 year
To ensure equivalent capecitabine exposure when compared to PK data from the same patients prior to gastrectomy. | 1 Year

CONTACTS AND LOCATIONS:
Overall Officials: Duncan Jodrell, DM MSc FRCP, Principal Investigator — Cambridge University Hospitals, NHS Foundation Trust, University of Cambridge
Locations (2):
- United Kingdom (2):
  - Cambridge University Hospitals NHS Foundation Trust, University of Cambridge Oncology Centre, Cambridge
  - Edinburgh Cancer Centre, Western General Hospital, Edinburgh